CLINICAL TRIAL: NCT02693912
Title: Changes in Alveolar Macrophage Function During Acute Lung Injury
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Chunling Jiang, Dr., West China Hospital
Other Study IDs: wch-150718
Record Dates: First submitted 2016-02-11; First posted 2016-02-29 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-02

CONDITIONS: Acute Lung Injury
Keywords: efferocytosis; macrophage
MeSH Terms: conditions — Acute Lung Injury | interventions — Bronchoscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — bronchoalveolar lavage fluid will be collected which contains immune cells, including macrophages.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- acute lung injury: Patients with a diagnosis of acute lung injury (ALI) under mechanical ventilation.Patients will underwent bronchoscopy for bronchoalveolar lavage fluid.
  Interventions: Procedure: Bronchoscopy
- control: Patient under mechanical ventilation without any lung diseases. Patients will underwent bronchoscopy for bronchoalveolar lavage fluid.
  Interventions: Procedure: Bronchoscopy

INTERVENTIONS:
Procedure: Bronchoscopy — Bronchoscopy will be implemented under sedation in both groups.

SUMMARY:
In this study, the investigators aim to observe the change in alveolar macrophage function during acute lung injury.

DETAILED DESCRIPTION:
Alveolar macrophages are tissue-resident or recruited cells with key functions in recognition of pathogens, initiation of host defensive ang protective inflammation,and in clearance of pathogens from the airways. However, macrophages are also responsible for efficient clearance of apoptotic neutrophils, termed efferocytosis, which is a prerequisite for the timely resolution of inflammation. In this study, the investigators aim to observe the change in alveolar macrophage function during acute lung injury.

ELIGIBILITY:
Inclusion Criteria:

* Patients in ICU with diagnosed ALI under mechanical ventilation

Exclusion Criteria:

* Patients with cardiac dysfunction, using steroid drugs or other drugs can that affect efferocytosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: ALI and acute respiratory distress syndrome (ARDS) are characterized by an increased permeability of the alveolar-capillary barrier resulting in lung edema with protein-rich fluid, thus resulting in impairment of arterial oxygenation. ALI/ARDS is defined as a lung disease with acute onset, noncardiac, diffuse bilateral pulmonary infiltrates and a paO2/FiO2 ≤ 300 for ALI or a paO2/FiO2 ≤ 200 for ARDS. The ageadjusted incidence of ALI/ARDS is estimated with 86.2 per 100,000 person-years. Despite all innovations in intensive care medicine, the mortality of ARDS remains up to 40%.
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-12 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
alveolar macrophages (AMs) phagocytic index | 7 days after admission
  AMs will be collected and cultured in vitro. Apoptotic neutrophils will then be cocultured with AMs for 1 hour. To measure phagocytosis of apoptotic neutrophils, AMs were further processed and phagocytosed apoptotic neutrophils were detected by confocal fluorescence microscopy as described below under Cell staining and confocal microscopy. The phagocytic index was calculated according to the following formula: phagocytic index = (total number of engulfed cells/total number of counted macrophages) × (number of macrophages containing engulfed cells/total number of counted macrophages) × 100.

SECONDARY OUTCOMES:
30 days mortality | 30 days after admission

CONTACTS AND LOCATIONS:
Overall Officials: Jin Liu, Study Chair — West China Hospital

IPD SHARING:
Plan to Share IPD: No
no plan has been made to share data